CLINICAL TRIAL: NCT03920397
Title: Allogenic Adipose Derived Mesenchymal Stem Cells and Vitamin D Supplementation in Patients With Recent-onset Type 1 Diabetes Mellitus
Brief Title: Mesenchymal Stem Cells in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Débora Lopes Souto, Ph. D. in Nutrition Sciences, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nutro_MesenchymalStemCells_DM1
Record Dates: First submitted 2019-04-05; First posted 2019-04-18 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; pancreatic function; adipose tissue-derived stromal/stem cells
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Patients with recent onset type 1 diabetes wil receive an dose of allogenic adipose tissue-derived stem/stromal cells (ASCs) and oral Cholecalciferol UI/day for 24 months.
Masking Description: This is a open trial study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose tissue-derived stem/stromal cells (Experimental): Safety of adipose tissue-derived stem/stromal cells (ASCs) for 24 months in patients with recente onset type 1 diabetes.
  Interventions: Biological: Infusion of adipose tissue-derived stem/stromal cells and oral Cholecalciferol supplementation
- Daily 2000 UI of daily oral cholecalciferol (Experimental): To investigate the efficacy of daily 2000 UI Cholecalciferol/day for 24 months in patients with recente onset type 1 diabetes.
  Interventions: Biological: Infusion of adipose tissue-derived stem/stromal cells and oral Cholecalciferol supplementation

INTERVENTIONS:
Biological: Infusion of adipose tissue-derived stem/stromal cells and oral Cholecalciferol supplementation — The investigators will acess area under the curve of C-peptide after a liquid mixed meal (Glucerna®), considering the time 0 (basal), 30, 60, 90 and 120 minutes in each follow-up outpatient visit (3 [T3], 6 [T6], 12 [T12], 18 [T18], and 24 [T24] months after the adipose tissue-derived stem/stromal cells infusion). Other Clinical and Pancreatic Function Evaluation that wil be assess are: Weight, height, body mass index (BMI), blood pressure, heart frequency, frequency of hypoglycemia and insulin dose/kg of body weight, blood count, lipids, renal and hepatic function, thyroid stimulating hormone, free tyroxine, antithyroglobulin antibody, calcium, phosphorus and 25-Hydroxy Vitamin D.

SUMMARY:
In this prospective, dual-center, open trial, patients with recent onset type 1 diabetes will receive one dose of allogenic Adipose tissue-derived stromal/stem cells (1x106 cells/kg) and oral cholecalciferol 2000UI/day for 24 months (group 1). They will be compare to patients that will receive just oral cholecalciferol 2000UI/day (group 2) and standard treatment (group 3: no treatment). Adverse events will be record. In addition, glycated hemoglobin, insulin dose, frequency of hypoglycemia, glycemic variability, % of time in hyper and hypoglycemia and peak response of the C-peptide after the mixed meal teste wil be measure at baseline (T0), after 3 (T3), 6 (T6), 12 (T12), 18 (T18), and 24 (T24) months.

DETAILED DESCRIPTION:
Adipose tissue samples will be obtain through liposuction procedures of three healthy volunteers undergoing aesthetic surgery at Clementino Fraga Filho (the hospital of Federal University of Rio de Janeiro, Brazil). Donors´sorology wil have to be negative for syphilis, Chagas disease, Hepatitis B virus, Hepatitis C, HIV 1 and 2, and Cytomegalovirus.

The adipose tissue-derived stem/stromal cells (ASCs) that wil be extract on healthy volunteers will be isolate, culture and samples will be process at Core Cell Technology of Pontifícia Universidade Católica do Paraná. Briefly, the procedures are:

1. 100 ml of adipose tissue will be wash in sterile phosphate-buffered saline (Gibco Invitrogen). A one-step digestion by 1 mg/ml collagenase type I (Invitrogen) will be performe for 30 minutes at 37°C during permanent shaking, follow by filtration step through a 100 µm mesh filter (BD FALCON, BD Biosciences Discovery Labware, Bedford, MA, USA). The cell suspension will be centrifuge at 800 g for 10 minutes, and erythrocytes were removed by lysis buffer, pH 7.3.
2. The remaining cells will be wash at 400 g for 10 minutes and then culture at a density of 1×105 cells/cm2 in T75 culture flasks and DMEM-F12 (Gibco Invitrogen) supplemente with 10% of fetal calf serum, penicillin (100 units/ml) and streptomycin (100 μg/ml). The culture medium will be replace three days after seeding, and then twice a week.
3. ASCs will be subculture after reaching 80% confluence, with 0.5% trypsin/EDTA (Invitrogen) solution. Cells will be replate at a density of 4x103 cells/cm2 for expansion11A.
4. Quality control of cell suspension sterility will be evaluate by tests to detect bacteria and fungi (Bact / Alert 3D, Biomerieux), endotoxins (Endosafe ™ PTS, Charles River) and Mycoplasma (KIT MycoAlert ™ PLUS Mycoplasma Detection, Lonza). Cell viability will be performe by flow cytometry using the vital dye 7-AAD (7-Aminoactinomycin D - BD#559925) to determine the percentage of viable cells and Annexin V protein (BD#51-65875X) to determine the percentage of cells in apoptosis. Cytogenetic analysis wil be performe by GTG-banding method.
5. Cells will be phenotypically characterize by flow cytometry before the clinical application, using the following monoclonal antibodies: FITC-labeled CD14 (BD#555397), CD45 (BD#555482), CD19 (BD#555412), CD44 (BD#555478); PE-labeled CD73 (BD#550257), CD90 (BD#555596), CD166 (BD#559263), PerCP-labeled HLA-DR (BD#551375); APC-labeled CD34 (BD#555824), CD105 (BD#562408), CD29 (BD#559883) all purchased from BD (Pharmingen). At least 100.000 events wil bel acquire on a BD FACSCalibur™ flow cytometer (BD Biosciences), and data wil be analyzed using FlowJo 10 (TreeStar) software11A.

After the ASCs extraction, isolate, culture and process, the infusion in patients with recent-onset type 1 diabetes wil be according as describe bellow:

1. At the day of infusion, ASCs monolayer wil be dissociate as described above and 1x106 cells/kg of the recipient patient wil be ressuspend in 5 ml of saline solution with 50% albumin and 5% anticoagulant citrate dextrose solution. Cell suspension wil send to the hospital in a cooler with recycled ice.
2. Patients that wil receive ASCs wil be admitte to the hospital in the day of the infusion and wil discharge 24 hours after infusion. A single dose of ASCs wil be infuse in a peripheral upper arm vein during 15-20 minutes. Patients wil start takking oral cholecalciferol 2000 UI one day after the ASCs infusion.

Safety Tests: adverse events wil be record during the hospitalization (T0) and at each follow-up outpatient visit (3 [T3], 6 [T6], 12 [T12], 18 [T18], and 24 [T24] months after the ASCs infusion), with clinical and laboratory exams (blood count, lipids, renal and hepatic function, thyroid stimulating hormone, free tyroxine, antithyroglobulin antibody, calcium, phosphorus and 25-Hydroxy Vitamin D, performed with automated biochemical equipment CMD 800 IX1).

Clinical and Pancreatic Function Evaluation: Participants wil be followed for 24 months. On the first visit, all patients wil be interviewed and had a physical exam. Weight, height, body mass index (BMI), blood pressure, heart frequency, frequency of hypoglycemia and insulin dose/kg of body weight wil be evaluate in the first visit (T0) and after 1 (T1), 3 (T3), 6 (T6) 12 (T12) ,18 (18), and 24 (24) months.

Insulin dose adjustments wil be performe at each visit as necessary. All patients wil receive nutritional guidance according to American Diabetes Association recommendations.

Blood samples wil be drawn prio to ASCs infusion and at T1, T3, T6, T12, T18 and T24 for the measurement the Glycated hemoglobin (HbA1c. Method: High Performance Liquid Chromatography by boronate affinity). β-cell function wil be evaluated through C-Peptide measurement (Microparticle Chemiluminescent Immunoassay method, Architect Abbott) after a liquid mixed meal (Glucerna®), considering the time 0 (basal), 30, 60, 90 and 120 minutes. The area under the curve wil be calculate.

Comparison with previous case-control study using only vitamin D supplementation as intervention:

The investigators wil compare our results with patients previously included in a case-control study that investigated the effects of daily 2000 UI vitamin D without the infusion of cells in individuals with recent onset type 1 diabetes and similar age (> 15 years old), from a different population (São Paulo) in the same country region (Brazilian Southeast). Therefore, the investigators wil establish three different groups for comparison: 1) patients that wil receive ASCs + Vitamin D supplementation; 2) patients that wil receive only vitamin D supplementation; 3) patients that wil receive the conventional treatment for diabetes but any additional experimental treament (ASCs or Vitamin D).

Insulin dose adjustments or withdrawal wil be performed according to glycemic control. Changes in HbA1c, C-Peptide and insulin dose/kg of body weight wil be compare between groups. C-Peptide wil be analyze by immunofluorometric assay (AutoDelfia) at T0 and T6 and T12 and T18 and T24, considering basal and peak stimulated C-Peptide after mixed meal test (Glucerna).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes according to the American Diabetes Association criteria for a period less than four months.
* Pancreatic Autoimmunity (positive anti-glutamic acid decarboxylase [GAD]; and/or Islet antigen 2 [anti-IA2]).

Exclusion Criteria:

* Clinical evidence of malignancy or prior history.
* Pregnancy or desire to become pregnant within 12 months of the study.
* Breastfeeding .
* HIV(+), Hepatitis B (+), Hepatitis C(+).
* Diabetic ketoacidosis at diagnosis.
* Glomerular filtration rate less than 60ml/min.
* Use of immunosuppressors or glucocorticoids.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Pancreatic β-cell function after an adipose tissue-derived stem/stromal cells infusion | 24 months
  Thirth patients with recent-onset type 1 diabetes wil receive adipose tissue-derived stem/stromal cells (ASCs). The patients wil be admitte in the day of the infusion and wil discharge 24 hours after infusion. A single dose of ASCs wil be infuse in a peripheral upper arm vein during 15-20 minutes.
  Pancreatic β-cell function will be assess at each follow-up outpatient visit (1, 3, 6, 12, 18 and 24 months after the ASCs infusion). In each visit, C-Peptide wil be analyze by immunofluorometric assay, considering the time 0 (basal), and peak stimulated C-Peptide (30, 60, 90 and 120 minutes) after mixed meal test (Glucerna)
Glycemic control after an adipose tissue-derived stem/stromal cells | 24 months
  Thirth patients with recent-onset type 1 diabetes wil receive adipose tissue-derived stem/stromal cells (ASCs). The patients wil be admitte in the day of the infusion and wil discharge 24 hours after infusion. A single dose of ASCs wil be infuse in a peripheral upper arm vein during 15-20 minutes.
  Frequency of hypoglycemia (%) insulin dose/kg, and blood samples will be drawn for the Glycated hemoglobin assessment (High Performance Liquid Chromatography by boronate affinity) at each follow-up outpatient visit (1, 3, 6, 12, 18 and 24 months after the ASCs infusion)

SECONDARY OUTCOMES:
Oral cholecalciferol 2000UI/day supplementation | 24 months
  The same patients with recent-onset type 1 diabetes wil receive adipose tissue-derived stem/stromal cells (ASCs) will receive Oral cholecalciferol 2000UI/day supplementation for 24 months.
  The sérum 25-Hydroxy Vitamin D will be assess at each follow-up outpatient visit (1, 3, 6, 12, 18 and 24 months after the ASCs infusion) and C-Peptide wil be analyze by immunofluorometric assay, considering the time 0 (basal), and peak stimulated C-Peptide (30, 60, 90 and 120 minutes) after mixed meal test (Glucerna)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Rodacki, Ph.D, Principal Investigator — Universidade Federal do Rio de Janeiro; Oliveira E.P José, Ph.D, Study Director — Universidade Federal do Rio de Janeiro; Lenita Zajdenverg, Ph.D, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Clementino Fraga Filho University Hospital of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dantas JR, Araujo DB, Silva KR, Souto DL, de Fatima Carvalho Pereira M, Luiz RR, Dos Santos Mantuano M, Claudio-da-Silva C, Gabbay MAL, Dib SA, Couri CEB, Maiolino A, Rebelatto CLK, Daga DR, Senegaglia AC, Brofman PRS, Baptista LS, de Oliveira JEP, Zajdenverg L, Rodacki M. Adipose tissue-derived stromal/stem cells + cholecalciferol: a pilot study in recent-onset type 1 diabetes patients. Arch Endocrinol Metab. 2021 Nov 3;65(3):342-351. doi: 10.20945/2359-3997000000368. Epub 2021 Apr 29. PMID 33939911
- [Derived] Araujo DB, Dantas JR, Silva KR, Souto DL, Pereira MFC, Moreira JP, Luiz RR, Claudio-Da-Silva CS, Gabbay MAL, Dib SA, Couri CEB, Maiolino A, Rebelatto CLK, Daga DR, Senegaglia AC, Brofman PRS, Baptista LS, Oliveira JEP, Zajdenverg L, Rodacki M. Allogenic Adipose Tissue-Derived Stromal/Stem Cells and Vitamin D Supplementation in Patients With Recent-Onset Type 1 Diabetes Mellitus: A 3-Month Follow-Up Pilot Study. Front Immunol. 2020 Jun 2;11:993. doi: 10.3389/fimmu.2020.00993. eCollection 2020. PMID 32582156